CLINICAL TRIAL: NCT03632512
Title: Effect of Hericium Erinaceus on Clinical Patients With Hearing Impairment and Possible Mechanisms
Brief Title: Effect of Hericium Erinaceus on Clinical Patients With Hearing Impairment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Providence University, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: B10604025
Record Dates: First submitted 2018-06-26; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Tinnitus
Keywords: Hericium erinaceus; Hearing
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hericium honey bolus (Experimental): Dosage form: honey bolus Dosage : Hericium erinaceus mycelium 250mg/day Frequency: 8 bolus/ day Duration: 8 months
  Interventions: Dietary Supplement: Hericium honey bolus
- Control group (Placebo Comparator): Dosage form: Placebo honey bolus Dosage : maize starch Frequency: 8 bolus/ day Duration: 8 months
  Interventions: Dietary Supplement: Placebo honey bolus

INTERVENTIONS:
Dietary Supplement: Hericium honey bolus — The subjects of the experimental group will be supplemented with Hericium Erinaceus honey bolus(430 mg/kg/day) for eight months.
  Arms: Hericium honey bolus
Dietary Supplement: Placebo honey bolus — The subjects of the control group will be supplemented with Placebo honey bolus(8 bolus/ day) for 8 months.
  Arms: Control group

SUMMARY:
This study aims to investigate the effect of Hericium Erinaceus on clinical patients with hearing impairment and possible mechanisms. Subjects with hearing impairment will be enrolled and randomly divided into experimental or control group supplemented with Hericium Erinaceus (430 mg/kg/day) or placebo, respectively for eight months. Basic characteristics will be evaluated at baseline by questionnaire. The hearing, liver and kidney functions, and neurotrophic factors will be examined at baseline, 4th month and 8th month.

DETAILED DESCRIPTION:
This study aims to investigate the effect of Hericium Erinaceus on clinical patients with hearing impairment and possible mechanisms. Subjects with hearing impairment will be enrolled. Inclusion criteria were 50 to 79 years old with symmetric sensorineural hearing loss, subjective sensorineural tinnitus, and all frequencies differed of ears less than 15 dB. Exclusion conditions were patients with abnormal liver and kidney function, normal hearing, severe and very severe hearing loss, no tinnitus or non-subjective sensorineural tinnitus, moderate or more cognitive impairment, patients unable to understand the details of this study or patients unable to co-examine, history of alcohol or drug abuse, history of high ambient noise exposure, bone tone air gap of pure tone hearing threshold greater than 10 dB, and audiogram 4 kHz air conduction threshold greater than 8 kHz, 20 dB airway threshold, hearing impairment before age 30, and inability to understand the details of this study. Participants will randomly divide into experimental or control group supplemented with Hericium Erinaceus (430 mg/kg/day) or placebo, respectively for eight months by a prospective, randomized, double-blind approach. Basic characteristics will be evaluated at baseline by questionnaire. The status of hearing, and CBC, GOT, GPT, BUN, Creatinine, NGF and BDNF expressions in blood will be examined at baseline, 4th month and 8th month.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 to 79 years old with symmetric sensorineural hearing loss, subjective sensorineural tinnitus, and all frequencies differed of ears less than 15 dB.

Exclusion Criteria:

* Patients with abnormal liver and kidney function, normal hearing, severe and very severe hearing loss, no tinnitus or non-subjective sensorineural tinnitus, moderate or more cognitive impairment , patients unable to understand the details of this study or patients unable to co-examine, history of alcohol or drug abuse, history of high ambient noise exposure, bone tone air gap of pure tone hearing threshold greater than 10 dB, and audiogram 4 kHz air conduction threshold greater than 8 kHz, 20 dB airway threshold, hearing impairment before age 30, and inability to understand the details of this study.

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-01-17 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
1.Change of Tinnitus status evaluates by Tinnitus handicap inventory (THI) | Baseline, 4th month and 8th month
  The status of tinnitus will be evaluated by Tinnitus handicap inventory (THI). THI is divided into three categories, including the functional (12 questions), emotional (8 questions), and catastrophic (5 questions) subscore. A total of 25 questions are used. The answer will be divided into three levels (will, sometimes, will not), and be scored into 4, 2 and 0 point, respectively. The subscore of functional (12 questions), emotional (8 questions), and catastrophic (5 questions) are 48, 32, and 20, respectively. The highest total score is 100 points. The higher the score, the more the tinnitus is. The difference of score will be compared from the baseline with 4th and 8th month.
Change of Tinnitus severity evaluates by visual analog scale (VAS) | Baseline, 4th month and 8th month
  The severity of tinnitus will be scored with a visual analog scale (VAS) from point 0 to point 10 by subject. The difference of score will be compared from the baseline with 4th and 8th month.
Changes of hearing obstacle average measure by Pure Tone Audiometry(PTA) | Baseline, 4th month and 8th month
  Pure tone threshold of subjects will be measured by Pure Tone Audiometry (PTA) to evaluate the changes from baseline ageing hearing obstacle average (dB HL) with 4th and 8th month.
Changes of speech recognizing measure by Speech Audiometry. | Baseline, 4th month and 8th month
  The Speech Audiometry is used to evaluate the changes of baseline speech recognizing (dB HL) and speech speech recognition rate(%) with 4th and 8th month.
Changes of NGF and BDNF levels of blood investigate by enzyme-linked immunosorbent assay (ELISA) | Baseline, 4th month and 8th month
  The NGF and BDNF levels of blood will be analyzed by enzyme-linked immunosorbent assay (ELISA) to detect the presence of NGF and BDNF. The NGF and BDN levels will be quantitative by the optical density (OD) of the sample comparing to a standard curve, which is a serial dilution of a known-concentration solution of the target molecule. The difference of NGF and BDNF levels will be compared from the baseline with 4th and 8th month.

CONTACTS AND LOCATIONS:
Overall Officials: Yin-Ching Chan, Study Chair — Providence University
Locations (1):
- Departments of Otolaryngology and Neurosurgery of Dalin Tzu Chi Hospital, Dalin, Chiayi, Taiwan

IPD SHARING:
Plan to Share IPD: No